CLINICAL TRIAL: NCT00946335
Title: A Phase I Study of ABT-888, an Oral Inhibitor of Poly (ADP-Ribose) Polymerase and Temozolomide in Children With Recurrent/Refractory CNS Tumors
Brief Title: ABT-888 and Temozolomide in Treating Young Patients With Recurrent or Refractory CNS Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03177; NCI-2012-03177 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR649727; PBTC-027 (Other: Pediatric Brain Tumor Consortium); PBTC-027 (Other: CTEP); U01CA081457 (NIH)
Record Dates: First submitted 2009-07-24; First posted 2009-07-27 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-06

CONDITIONS: Childhood Atypical Teratoid/Rhabdoid Tumor; Childhood Central Nervous System Germ Cell Tumor; Childhood Choroid Plexus Tumor; Childhood Craniopharyngioma; Childhood Ependymoblastoma; Childhood Grade I Meningioma; Childhood Grade II Meningioma; Childhood Grade III Meningioma; Childhood High-grade Cerebellar Astrocytoma; Childhood High-grade Cerebral Astrocytoma; Childhood Infratentorial Ependymoma; Childhood Low-grade Cerebellar Astrocytoma; Childhood Low-grade Cerebral Astrocytoma; Childhood Medulloepithelioma; Childhood Mixed Glioma; Childhood Oligodendroglioma; Childhood Supratentorial Ependymoma; Recurrent Childhood Brain Stem Glioma; Recurrent Childhood Brain Tumor; Recurrent Childhood Cerebellar Astrocytoma; Recurrent Childhood Cerebral Astrocytoma; Recurrent Childhood Ependymoma; Recurrent Childhood Medulloblastoma; Recurrent Childhood Pineoblastoma; Recurrent Childhood Spinal Cord Neoplasm; Recurrent Childhood Subependymal Giant Cell Astrocytoma; Recurrent Childhood Supratentorial Primitive Neuroectodermal Tumor; Recurrent Childhood Visual Pathway and Hypothalamic Glioma
MeSH Terms: conditions — Rhabdoid Tumor; Choroid Plexus Neoplasms; Astrocytoma; Oligodendroglioma; Familial ependymoma; Medulloblastoma; Spinal Cord Neoplasms; Optic Nerve Glioma | interventions — veliparib; Temozolomide

ARMS (1):
- Treatment (veliparib, temozolomide) (Experimental): Patients receive oral ABT-888 twice daily and oral temozolomide once daily on days 1-5. Treatment repeats every 28 days for 13-26 courses in the absence of disease progression or unacceptable toxicity.
  Blood samples are collected for pharmacokinetics and further laboratory analysis.
  Interventions: Drug: veliparib; Drug: temozolomide; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: veliparib — Given PO
  Other Names: ABT-888
Drug: temozolomide — Given PO
  Other Names: SCH 52365; Temodal; Temodar; TMZ
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial is studying the side effects and best dose of ABT-888 when given in combination with temozolomide in treating young patients with recurrent or refractory CNS tumors. ABT-888 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving ABT-888 together with temozolomide may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the maximum tolerated dose (MTD) of ABT-888 in combination with temozolomide in children with recurrent or refractory CNS tumors.

II. To study the plasma pharmacokinetics (PK) of ABT-888 and PARP inhibition in peripheral blood mononuclear cells (PBMC) in order to recommend a Phase 2 dose of ABT-888 in combination with temozolomide in children with recurrent or refractory CNS tumors.

III. To describe the toxicities of the combination of ABT-888 and temozolomide in children with recurrent or refractory CNS tumors.

SECONDARY OBJECTIVES:

I. To measure non-homologous end-joining (NHEJ) activity in peripheral blood mononuclear cells (PBMC) prior to and following ABT-888 administration.

II. To assess PARP expression and/or activity in tumor tissue obtained at either initial diagnosis or relapse.

III. To determine expression and/or activity of DNA repair pathways, including MGMT and mismatch repair, in tumor tissues, when available.

IV. To document, within the confines of this phase 1 trial, radiographic tumor response to ABT-888 and temozolomide.

OUTLINE: This is a dose-escalation study of ABT-888.

Patients receive oral ABT-888 twice daily and oral temozolomide once daily on days 1-5. Treatment repeats every 28 days for 13-26 courses in the absence of disease progression or unacceptable toxicity.

Blood samples are collected for pharmacokinetics and further laboratory analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of a primary CNS malignancy (including low-grade glioma) that is recurrent or refractory to standard therapy and for which there is no known curative therapy; all patients must have had histological verification of malignancy at initial diagnosis or relapse, excluding patients with diffuse intrinsic brain stem tumors, optic pathway tumors or CNS germ cell tumors with elevations of reliable serum or CSF tumor markers (alpha-fetoprotein or beta-HCG); patients with intrinsic pontine gliomas or optic pathway tumors do not require histological confirmation of disease but should have clinical and/or radiographic evidence of progression
* Patients must have Karnofsky Performance Score (for patients > 16 years of age) or Lansky Performance Score (for patients =< 16 years of age) >= 50% assessed within two weeks of study enrollment
* Patients must be able to take oral medications (either capsules or liquid); patients with neurologic deficits must have been stable for a minimum of 1 week prior to study entry; patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study; recovery is defined as all AE"s, attributable to prior therapy, having improved to grade 2 or better or as outlined below
* Myelosuppressive chemotherapy:

  * Patients must have received their last dose of known myelosuppressive anticancer chemotherapy at least three (3) weeks prior to study registration
  * Patients must have received their last dose of nitrosourea (including Gliadel) at least six (6) weeks prior to study registration
* Biologic agent (anti-neoplastic): Patient must have received their last dose of other biologic agent ≥ 7 days prior to study registration

  * For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur; the duration of this interval must be discussed with the study chair
* Monoclonal antibody treatment: Patient must have received their last dose of monoclonal antibody ≥ 4 weeks prior to registration
* Radiation - Patients who have had prior radiation must have had their last fraction of:

  * Craniospinal irradiation or total body irradiation > 3 months prior to registration
  * Local irradiation to the primary tumors or other sites (cumulative dose ≥ 40Gy) > 3 months prior to registration
  * Palliative irradiation delivered to symptomatic metastatic sites > 4 weeks prior to registration
* Stem Cell Transplant: Patient must be:

  * ≥ 6 months since allogeneic stem cell transplant prior to registration
  * ≥ 3 months since autologous stem cell transplant prior to registration
* Corticosteroids: Patients who are receiving dexamethasone must be on a stable or decreasing dose for at least 1 week prior to registration
* Growth factors:

  * Off all colony forming growth factor(s) that support platelet or white blood cell count, number or function for at least 1 week prior to registration (filgrastim, sargramostim, erythropoietin)
  * Off Pegylated G-CSF and/or Erythropoiesis Stimulating Protein for at least 14 days prior to registration
* Temozolomide: Patients who have received temozolomide previously are eligible for this study if they meet all other inclusion and exclusion criteria
* Organ Function: Documented within 14 days of registration and within 7 days of starting treatment
* Hgb > 8 gm/dL (transfusion independent)
* Platelet count > 100,000/mm^3 (transfusion independent)
* Absolute neutrophil count (ANC) > 1, 500/mm^3
* Total Bilirubin (sum of conjugated + unconjugated) ≤ 1.5 times institutional upper limit of normal (ULN) for age
* SGPT (ALT) ≤ 2.5 times institutional ULN for age
* Serum albumin ≥ 2 g/dL
* Creatinine clearance or radioisotope GFR ≥ 70 ml/min/1.73m^2 or a serum creatinine based on age as follows:

  * ≤ 5 years - 0.8 mg/dL maximum serum creatinine
  * > 5 to ≤ 10 years - 1 mg/dL maximum serum creatinine
  * > 10 to ≤ 15 years - 1.2 mg/dL maximum serum creatinine
  * > 15 years - 1.5 maximum serum creatinine
* Patients must not be pregnant or breast-feeding; females of reproductive potential must have a negative serum or urine pregnancy test (within 72 hours prior to enrollment); males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method, which includes abstinence
* Signed informed consent which includes consent to participate in the REQUIRED pharmacokinetic and pharmacodynamic studies prior to registration

Exclusion Criteria:

* Patients receiving any of the following medications are not eligible for study entry:

  * Anti-cancer therapy
  * Investigational agents
* Patients with any clinically significant, unrelated systemic illness (serious infections or significant cardiac, pulmonary, hepatic or other organ dysfunction), that would compromise the patient's ability to tolerate protocol therapy or would likely interfere with the study procedures or results
* Patients with uncontrolled seizures are not eligible for study entry
* Patients with inadequately controlled systemic hypertension (SBP and/or DBP > 95th percentile for age and height
* Patients with a prior history of hypertensive crisis and/or hypertensive encephalopathy
* If a BP measurement prior to registration is > 95th percentile for age and height, it must be rechecked and documented to be < 95th percentile for age and height prior to registration; if a patient falls between the height or weight percentiles, site should average the value as appropriate; for patients ≥ 18 years the normal blood pressure should be < 140/90 mm of Hg; patients with hypertension are eligible if their blood pressures become < 95th percentile for age and height after anti-hypertensive medications
* Patients with documented CNS ischemia and/or infarction, whether symptomatic or discovered incidentally without clinical symptoms, will be excluded from study participation
* Patients with an inability to return for follow-up visits or obtain follow-up studies required to assess toxicity to therapy

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2009-07; Primary Completion 2011-10 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
MTD or recommended phase II dose of veliparib | 28 days
Acute toxicities | Initial 4 weeks (course 1)
  These toxicities will be tabulated according to dose level.
Chronic toxicities | Up to 30 days post-treatment
  Tabulated according to dose level and course of therapy.
Plasma drug concentrations and pharmacokinetic parameters, including volume of the central compartment (Vc/F), elimination rate constant (Ke), half-life (t1/2), apparent oral clearance (CL/F), and area under the plasma concentration time curve (AUC) | Baseline and during course 1
  Presented in tabular and graphical form, and estimated using compartmental methods. Dose proportionality in pharmacokinetic parameters will be investigated by performing one-way analysis of variance (ANOVA) on dose-normalized parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Jack Su, Principal Investigator — Pediatric Brain Tumor Consortium
Locations (1):
- Pediatric Brain Tumor Consortium, Memphis, Tennessee, United States